CLINICAL TRIAL: NCT06821906
Title: Stereotactic Radiosurgery in the Treatment of Tremor in Patients with Essential Tremor - a Randomized Phase II Study
Brief Title: Stereotactic Radiosurgery in the Treatment of Essential Tremor
Acronym: EASIER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EASIER
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Essential Tremor
Keywords: tremor; stereotactic radiosurgery; frameless radiosurgery; essenstial tremor; CyberKnife
MeSH Terms: conditions — Essential Tremor; Tremor | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Randomised, open label, interventional research experiment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Active Comparator): Patients irradiated with the CyberKnife with a dose of 130 Gy
  Interventions: Radiation: Stereotactic Radiosurgery
- B (Experimental): Patients irradiated with the CyberKnife with a dose of 80 Gy
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Frameless Stereotactic Radiosurgery- CyberKnife with a dose of 80 Gy
  Arms: B
Radiation: Stereotactic Radiosurgery — Frameless Stereotactic Radiosurgery- CyberKnife with a dose of 130 Gy
  Arms: A

SUMMARY:
The goal of this interventional study is to evaluate the effectiveness of treatment using stereotactic radiosurgery in the treatment of essential tremor in adult patients

DETAILED DESCRIPTION:
The study will include patients diagnosed with essential tremor who have insufficient tremor control despite the use of available pharmacotherapy methods. The study will include patients who have been disqualified from the Deeply Brain Stimulation procedure or who do not consent to its performance. Additional conditions for the examination are age over 50 and the duration of the disease over 5 years.

After qualifying and giving written informed consent, the patient will be randomly assigned to one of two study arms:

1. control arm: patients irradiated with the CyberKnife with a dose of 130 Gy
2. test arm: patients irradiated with the CyberKnife with a dose of 80 Gy

The primary aim of the study is to determine the effectiveness of radiosurgery in patients with essential tremor. Secondary objectives will be to determine the impact of treatment on the quality of life of, as well as to assess the safety and possible complications of radiosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Essential tremor diagnosed, Parkinson's disease and other causes of tremor excluded.
* Insufficient tremor control despite the use of available pharmacotherapy methods.
* Disqualification from the Deeply Brain Stimualtion procedure/lack of consent to perform it on the side qualified for Stereotactic Radiosurgery
* Consent to participate in a clinical trial.

Exclusion Criteria:

* Age under 50
* Pregnancy
* Duration of the disease less than 5 years
* Dementia, psychosis or other condition that prevents giving informed consent to participate in the study
* Poor general condition, serious comorbidities
* Structural changes in the basal ganglia or major atrophic changes
* Previous radiotherapy to the brain covering the potential treatment area
* Medical contraindications to magnetic resonance imaging

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Treatment Efficacy | 24 months
  Efficacy of radiosurgery treatment in patients with essential tremor assessed on a dedicated tremor severity scale - Fahn-Tolosa-Marin (FTM)

SECONDARY OUTCOMES:
Quality of life | 24 months
  The impact of treatment on the quality of life of patients based on the dedicated Quality of Life in Essential Tremor questionnaire
Safety | 24 months
  Safety and possible complications of radiosurgery assesed in Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Napieralska, Principal Investigator — Maria Skłodowska-Curie National Research Institute of Oncology, Gliwice Branch
Locations (1):
- Maria Skłodowska-Curie National Research Institute of Oncology, Gliwice Branch, Gliwice, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Louis ED, Ferreira JJ. How common is the most common adult movement disorder? Update on the worldwide prevalence of essential tremor. Mov Disord. 2010 Apr 15;25(5):534-41. doi: 10.1002/mds.22838. PMID 20175185
- [Background] Bhatia KP, Bain P, Bajaj N, Elble RJ, Hallett M, Louis ED, Raethjen J, Stamelou M, Testa CM, Deuschl G; Tremor Task Force of the International Parkinson and Movement Disorder Society. Consensus Statement on the classification of tremors. from the task force on tremor of the International Parkinson and Movement Disorder Society. Mov Disord. 2018 Jan;33(1):75-87. doi: 10.1002/mds.27121. Epub 2017 Nov 30. PMID 29193359
- [Background] Hopfner F, Haubenberger D, Galpern WR, Gwinn K, Van't Veer A, White S, Bhatia K, Adler CH, Eidelberg D, Ondo W, Stebbins GT, Tanner CM, Helmich RC, Lenz FA, Sillitoe RV, Vaillancourt D, Vitek JL, Louis ED, Shill HA, Frosch MP, Foroud T, Kuhlenbaumer G, Singleton A, Testa CM, Hallett M, Elble R, Deuschl G. Knowledge gaps and research recommendations for essential tremor. Parkinsonism Relat Disord. 2016 Dec;33:27-35. doi: 10.1016/j.parkreldis.2016.10.002. Epub 2016 Oct 4. PMID 27769649
- [Background] Jackson AL, Murphy LL. Role of the hypothalamic-pituitary-adrenal axis in the suppression of luteinizing hormone release by delta-9-tetrahydrocannabinol. Neuroendocrinology. 1997 Jun;65(6):446-52. doi: 10.1159/000127208. PMID 9208407
- [Background] Hooper AK, Okun MS, Foote KD, Fernandez HH, Jacobson C, Zeilman P, Romrell J, Rodriguez RL. Clinical cases where lesion therapy was chosen over deep brain stimulation. Stereotact Funct Neurosurg. 2008;86(3):147-52. doi: 10.1159/000120426. Epub 2008 Mar 12. PMID 18334856
- [Background] Niranjan A, Jawahar A, Kondziolka D, Lunsford LD. A comparison of surgical approaches for the management of tremor: radiofrequency thalamotomy, gamma knife thalamotomy and thalamic stimulation. Stereotact Funct Neurosurg. 1999;72(2-4):178-84. doi: 10.1159/000029723. PMID 10853075
- [Background] Young RF, Shumway-Cook A, Vermeulen SS, Grimm P, Blasko J, Posewitz A, Burkhart WA, Goiney RC. Gamma knife radiosurgery as a lesioning technique in movement disorder surgery. J Neurosurg. 1998 Aug;89(2):183-93. doi: 10.3171/jns.1998.89.2.0183. PMID 9688111
- [Background] Stancanello J, Romanelli P, Pantelis E, Sebastiano F, Modugno N. Atlas-based functional radiosurgery: early results. Med Phys. 2009 Feb;36(2):457-63. doi: 10.1118/1.3056460. PMID 19291984
- [Background] Bretsztajn L, Gedroyc W. Brain-focussed ultrasound: what's the "FUS" all about? A review of current and emerging neurological applications. Br J Radiol. 2018 Jul;91(1087):20170481. doi: 10.1259/bjr.20170481. Epub 2018 Mar 6. PMID 29419328
- [Background] LEKSELL L. The stereotaxic method and radiosurgery of the brain. Acta Chir Scand. 1951 Dec 13;102(4):316-9. No abstract available. PMID 14914373
- [Background] Lindquist C, Kihlstrom L, Hellstrand E. Functional neurosurgery--a future for the gamma knife? Stereotact Funct Neurosurg. 1991;57(1-2):72-81. doi: 10.1159/000099557. PMID 1725560
- [Background] Martinez-Moreno NE, Sahgal A, De Salles A, Hayashi M, Levivier M, Ma L, Paddick I, Regis J, Ryu S, Slotman BJ, Martinez-Alvarez R. Stereotactic radiosurgery for tremor: systematic review. J Neurosurg. 2018 Feb 23;130(2):589-600. doi: 10.3171/2017.8.JNS17749. Print 2019 Feb 1. PMID 29473775
- [Background] Duma CM. Movement disorder radiosurgery--planning, physics and complication avoidance. Prog Neurol Surg. 2007;20:249-266. doi: 10.1159/000100168. PMID 17317994
- [Background] Khattab MH, Cmelak AJ, Sherry AD, Luo G, Wang L, Yu H, Hedera P, Phibbs FT, Lindsell CJ, Neimat J, Kirschner AN. Noninvasive Thalamotomy for Refractory Tremor by Frameless Radiosurgery. Int J Radiat Oncol Biol Phys. 2022 Jan 1;112(1):121-130. doi: 10.1016/j.ijrobp.2021.08.021. Epub 2021 Aug 25. PMID 34454047
- [Background] Kim W, Sharim J, Tenn S, Kaprealian T, Bordelon Y, Agazaryan N, Pouratian N. Diffusion tractography imaging-guided frameless linear accelerator stereotactic radiosurgical thalamotomy for tremor: case report. J Neurosurg. 2018 Jan;128(1):215-221. doi: 10.3171/2016.10.JNS161603. Epub 2017 Feb 24. PMID 28298033
- [Background] Franzini A, Marchetti M, Brait L, Milanesi I, Messina G, Forapani E, Broggi G, Fariselli L. Deep brain stimulation and frameless stereotactic radiosurgery in the treatment of bilateral parkinsonian tremor: target selection and case report of two patients. Acta Neurochir (Wien). 2011 May;153(5):1069-75. doi: 10.1007/s00701-011-0962-0. Epub 2011 Feb 20. PMID 21336920
- [Background] Goc B, Roch-Zniszczol A, Larysz D, Zarudzki L, Stapor-Fudzinska M, Rozek A, Wozniak G, Boczarska-Jedynak M, Miszczyk L, Napieralska A. The Effectiveness and Toxicity of Frameless CyberKnife Based Radiosurgery for Parkinson's Disease-Phase II Study. Biomedicines. 2023 Jan 20;11(2):288. doi: 10.3390/biomedicines11020288. PMID 36830825
- [Background] Solberg TD, Medin PM, Mullins J, Li S. Quality assurance of immobilization and target localization systems for frameless stereotactic cranial and extracranial hypofractionated radiotherapy. Int J Radiat Oncol Biol Phys. 2008;71(1 Suppl):S131-5. doi: 10.1016/j.ijrobp.2007.05.097. PMID 18406912
- [Background] Luo G, Neimat JS, Cmelak A, Kirschner AN, Attia A, Morales-Paliza M, Ding GX. Margin of error for a frameless image guided radiosurgery system: Direct confirmation based on posttreatment MRI scans. Pract Radiat Oncol. 2017 May-Jun;7(3):e223-e231. doi: 10.1016/j.prro.2016.08.006. Epub 2016 Aug 20. PMID 27720703
- [Background] Yu C, Main W, Taylor D, Kuduvalli G, Apuzzo ML, Adler JR Jr. An anthropomorphic phantom study of the accuracy of Cyberknife spinal radiosurgery. Neurosurgery. 2004 Nov;55(5):1138-49. doi: 10.1227/01.neu.0000141080.54647.11. PMID 15509320
- [Background] Campbell AM, Glover J, Chiang VL, Gerrard J, Yu JB. Gamma knife stereotactic radiosurgical thalamotomy for intractable tremor: a systematic review of the literature. Radiother Oncol. 2015 Mar;114(3):296-301. doi: 10.1016/j.radonc.2015.01.013. Epub 2015 Feb 14. PMID 25690750
- [Background] Hashim M, Vincken T, Kroi F, Gebregergish S, Spencer M, Wang J, Kampfenkel T, Lam A, He J. A systematic review of noninferiority margins in oncology clinical trials. J Comp Eff Res. 2021 Apr;10(6):443-455. doi: 10.2217/cer-2020-0200. Epub 2021 Mar 17. PMID 33728935
- [Background] Palesch YY. Some common misperceptions about P values. Stroke. 2014 Dec;45(12):e244-6. doi: 10.1161/STROKEAHA.114.006138. Epub 2014 Nov 6. No abstract available. PMID 25378423
- [Background] Chow S-C., Shao J., Wang H., Lokhnygina Y. Sample Size Calculations in Clinical Research. Third ed: Chapman and Hall/CRC; 2017.